CLINICAL TRIAL: NCT00857701
Title: Dynamic Splinting After Total Knee Arthroplasty: a Randomized, Controlled Trial
Brief Title: Dynamic Splinting After Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unrelated to trial
Sponsor: Dynasplint Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008.009
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Reduced Knee Flexion
Keywords: total knee arthroplasty; Dynamic Splinting; Knee extension; knee; Reduced knee flexion after total knee arthroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Patient will receive post-surgical standard of care treatment with standard Physical therapy and NSAIDs.
- 2 (Experimental): Patients will be treated with the Standard of Care physical therapy and NSAIDs as well as a Knee Extension Dynasplint that includes tension chambers.
  Interventions: Device: Knee Extension Dynasplint

INTERVENTIONS:
Device: Knee Extension Dynasplint — Dynamic Splinting utilizes the protocols of Low-Load, Prolonged-Duration Stretch (LLPS) with calibrated, adjustable tension to increase the Total End Range Time (TERT) to reduce contracture. The Knee Extension Dynasplint for the Experimental group will have tension chambers delivering therapeutic treatment from the device.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a dynamic splinting system for knee flexion contracture following a total knee arthroplasty.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy of dynamic splinting for knee flexion contracture following a total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Reduced flexibility in AROM of knee extension
* Pain that is worsened by bending over while legs are straight
* Impaired gait pattern
* Ability to understand informed consent and experiment responsibilities

Exclusion Criteria:

* Fractures
* Knee sepsis
* Osteomyelitis or any orthopedic infection
* Extensor mechanism dysfunction
* Psoriasis
* Knee joint neuropathy
* Previous Stroke or Brain Injury

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-01; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Change in Maximal Acitive Range of Mothion in knee extension | 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dennis L Armstrong M.D., Mesa, Arizona, United States

REFERENCES:
- [Background] Denis M, Moffet H, Caron F, Ouellet D, Paquet J, Nolet L. Effectiveness of continuous passive motion and conventional physical therapy after total knee arthroplasty: a randomized clinical trial. Phys Ther. 2006 Feb;86(2):174-85. PMID 16445331
- [Background] Scuderi GR, Kochhar T. Management of flexion contracture in total knee arthroplasty. J Arthroplasty. 2007 Jun;22(4 Suppl 1):20-4. doi: 10.1016/j.arth.2006.12.110. PMID 17570272
- [Background] Kotani A, Yonekura A, Bourne RB. Factors influencing range of motion after contemporary total knee arthroplasty. J Arthroplasty. 2005 Oct;20(7):850-6. doi: 10.1016/j.arth.2004.12.051. PMID 16230234
- [Background] Jansen CM, Windau JE, Bonutti PM, Brillhart MV. Treatment of a knee contracture using a knee orthosis incorporating stress-relaxation techniques. Phys Ther. 1996 Feb;76(2):182-6. doi: 10.1093/ptj/76.2.182. PMID 8592722
- [Background] Fitzgerald GK, Childs JD, Ridge TM, Irrgang JJ. Agility and perturbation training for a physically active individual with knee osteoarthritis. Phys Ther. 2002 Apr;82(4):372-82. PMID 11922853
- [Background] Laskin RS, Beksac B. Stiffness after total knee arthroplasty. J Arthroplasty. 2004 Jun;19(4 Suppl 1):41-6. doi: 10.1016/j.arth.2004.02.008. PMID 15190548
- [Background] Bourne RB, Laskin RS, Guerin JS. Ten-year results of the first 100 Genesis II total knee replacement procedures. Orthopedics. 2007 Aug;30(8 Suppl):83-5. PMID 17824343
- [Background] Bradbury N, Borton D, Spoo G, Cross MJ. Participation in sports after total knee replacement. Am J Sports Med. 1998 Jul-Aug;26(4):530-5. doi: 10.1177/03635465980260041001. PMID 9689373
- [Background] Cloutier JM, Sabouret P, Deghrar A. Total knee arthroplasty with retention of both cruciate ligaments. A nine to eleven-year follow-up study. J Bone Joint Surg Am. 1999 May;81(5):697-702. doi: 10.2106/00004623-199905000-00011. PMID 10360698
- [Background] Kawamura H, Bourne RB. Factors affecting range of flexion after total knee arthroplasty. J Orthop Sci. 2001;6(3):248-52. doi: 10.1007/s007760100043. PMID 11484119
- [Background] Kahle JT, Highsmith MJ, Hubbard SL. Comparison of nonmicroprocessor knee mechanism versus C-Leg on Prosthesis Evaluation Questionnaire, stumbles, falls, walking tests, stair descent, and knee preference. J Rehabil Res Dev. 2008;45(1):1-14. doi: 10.1682/jrrd.2007.04.0054. PMID 18566922